CLINICAL TRIAL: NCT02183753
Title: Effects of Wood Smoke Particles on Influenza-induced Nasal Inflammation in Normal Volunteers
Acronym: Woodsies
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 13-3076; 5R01ES013611-09 (NIH)
Record Dates: First submitted 2014-06-03; First posted 2014-07-08 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Response of Viral Infection to Woodsmoke
Keywords: LAIV; Flumist; wood smoke
MeSH Terms: conditions — Influenza, Human | interventions — Environment, Controlled

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wood smoke (Active Comparator): The dose of WSP to be used (500 µg/m3 for 2 hours) is based on prior studies which indicate the exposure is well tolerated, and is similar to that found in some indoor exposures in homes heated by wood burning (24-26). The route of administration (breathing air containing WSP at rest, nasally) is intended to mimic natural exposures.
  Interventions: Other: wood smoke
- clean air (Placebo Comparator): Chapel Hill air which has been filtered to remove ambient air pollutants.
  Interventions: Other: clean air

INTERVENTIONS:
Other: wood smoke
  Arms: Wood smoke
Other: clean air
  Arms: clean air

SUMMARY:
This study is focused on the pathophysiology underlying the association between exposure to particulate pollutants and risk for/response to viral infection. The investigators hypothesize that exposure to wood smoke particles (WSP) enhances influenza virus-induced granulocyte and NK cell activation, via hyaluronic acid-mediated effects on IFNg production. Oxidant stress and viral replication may also be affected. As an NIH funded ViCTER project, the purpose of the study is also to test novel assays of granulocyte activation (Doershuk lab) and lipid mediator activation (Albritton lab) which have not previously been used in this type of research.

Healthy, nonsmoking adults age 18-40 years will be recruited. This is a randomized, placebo controlled study comparing NLF granulocyte responses to LAIV administered after either WSP or clean air, in normal healthy volunteers. Subjects receive either WSP or placebo (clean air), followed by a standardized dose of LAIV and serial post-infection sampling of nasal lavage fluids, nasal biopsy and blood

ELIGIBILITY:
Inclusion Criteria:

1. Normal lung function, defined as (Knudson 1976/1984 predicted set): FVC > 75 % predicted for gender, ethnicity, age and height; FEV1 >75 % predicted ; FEV1/FVC ratio >0.70 and < 0.90.
2. Oxygen saturation of > 94%
3. Normal blood pressure (Systolic between 140 - 90, Diastolic between 90-60 mm Hg)
4. Symptom Score no greater than 6 (out of a possible 39) for total symptom score
5. On the day of a challenge, body temperature must be no greater than 37.8 degrees, measured orally

Exclusion Criteria:

1. A history of significant chronic illnesses (to include diabetes, autoimmune diseases, immunodeficiency state, known ischemic heart disease, chronic respiratory diseases such as chronic obstructive pulmonary disease or asthma, hypertension)
2. Positive pregnancy test within 48 hours of the time of challenge
3. Use of any inhaled substance (for medical or recreational purposes). Nonsmokers must have been abstinent from smoking for the prior 12 months, having not smoked more than 1 pack over the course of the previous year and does not smoke at all 1 week prior to entrance in the study.
4. Receipt of LAIV in the current season
5. History of allergy to eggs
6. Acute, non-chronic, medical conditions, including (but not limited to) pneumonia or bronchitis requiring antibiotics, febrile illnesses, flu-like symptoms must be totally resolved symptomatically for 3 weeks
7. Unspecified illnesses, which in the judgment of the investigator increase the risk associated with the experimental LAIV infection, will be a basis for exclusion.
8. Expected exposure of subject to immunocompromised individuals (who can be infected by LAIV) for the 3 weeks following LAIV inoculation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
IL-13 | 1-21 days
  Change in IL-13 and ECP in nasal lavage fluids (NLF) compared to pre-virus baseline

CONTACTS AND LOCATIONS:
Overall Officials: Terry Noah, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- center for envionmental medicine asthma an lung biology at the EPA, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Rebuli ME, Speen AM, Martin EM, Addo KA, Pawlak EA, Glista-Baker E, Robinette C, Zhou H, Noah TL, Jaspers I. Wood Smoke Exposure Alters Human Inflammatory Responses to Viral Infection in a Sex-Specific Manner. A Randomized, Placebo-controlled Study. Am J Respir Crit Care Med. 2019 Apr 15;199(8):996-1007. doi: 10.1164/rccm.201807-1287OC. PMID 30360637